CLINICAL TRIAL: NCT01391429
Title: Testing a Video Decision Support Tool to Supplement Goals-of-Care Discussions With Patients and Surrogates Receiving an Inpatient Palliative Care Consult
Brief Title: Testing a Video Decision Support Tool to Supplement Goals-of-Care Discussions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Michael Paasche-Orlow, BMC Attending Physician, Boston Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H29666
Record Dates: First submitted 2011-06-21; First posted 2011-07-12 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Advance Care Planning; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video decision support tool (Experimental): Video decision support tool for goals-of-care options
  Interventions: Behavioral: Video Decision Support Tool
- Verbal description (No Intervention): Standard verbal description of goals-of-care options provided by an inpatient palliative care team

INTERVENTIONS:
Behavioral: Video Decision Support Tool — Six minute digital video illustrating specific treatments for three different levels of medical care: life-prolonging care, basic care and comfort oriented care.
  Arms: Video decision support tool

SUMMARY:
Subject preferences for care at the end-of-life show wide variability. In the setting of advanced disease, some subjects prefer all life-sustaining care while others forgo such procedures. The wide variability in preferences may be due to subjects' misconception of the disease condition when using solely verbal descriptions. The failure to participate in effective goals-of-care discussions may lead to overuse of medical interventions and life-sustaining measures that are inconsistent with patients' and families' wishes. Using video images -- in addition to words -- to convey goals-of-care options at end-of-life, adds a sense of verisimilitude to the condition described and may better inform subjects when making their preferences.

Specific Aim: To assess the effect of a video decision support tool on preferences for end-of-life care in patients and surrogate decision makers consulted on by an inpatient palliative care service. The investigators hypothesize that those subjects who view video images as a supplement to a standard palliative care consult will be more likely to opt for comfort oriented care.

In this study, patient subjects and/or their healthcare proxies who are consulted on by an inpatient palliative care team will be surveyed regarding their preferences for end-of-life care following either a standard palliative care consult or one which utilizes a short video to complement verbal descriptions. The primary analysis will involve the proportion of patient subjects/proxies in each group that prefer comfort oriented care and that die in accordance with their stated preferences. The investigators will also study the effect of the video on patient subjects' and/or proxies' uncertainty with regard to treatment preferences and overall satisfaction with the palliative care consult.

DETAILED DESCRIPTION:
The investigators research will be conducted as a non-randomized, temporal intervention study. The specific aim of the study is to assess the effect of a video decision support tool on preferences for end-of-life care in patients and surrogate decision makers consulted on by an inpatient palliative care service. The first seven months of the study, or until 25 patient subjects are recruited, will be the observational phase. All participants recruited will receive the usual standard of care provided by an inpatient palliative care service. Using a battery of surveys, data will be collected regarding treatment preferences near the end of life, level of certainty with decision making, pain and symptom management, resource utilization and whether patient subjects die in accordance with their stated preferences. Once the observational phase is complete, the intervention phase of the study will begin. Over the following seven months, or until 25 patient subjects are recruited, all participants will view a six-minute digital video outlining different options for care near the end of life. The same endpoints will then be followed. In addition to the primary analysis involving patient-proxy dyads, an additional exploratory analysis will be performed. This analysis will involve surveying additional medical staff including attendings, residents, interns and nurses regarding their perceptions of patients' symptoms at the time of the palliative care consult. This data will be used to measure concordance between patient subjects' and staffs' ranking of symptoms.

ELIGIBILITY:
Inclusion Criteria-patient subjects/proxies:

* Adult patients and their healthcare proxies consulted on by an inpatient palliative care team.
* English-speaking
* Potential patient subjects and/or their healthcare proxies must have the ability to provide informed consent.

Inclusion Criteria-staff subjects:

* Must be members of the palliative care or primary medical team

Exclusion Criteria:

* Potential patient subjects who are identified by the palliative care team as not being appropriate for a goals-of-care discussion will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The difference in proportions of patient subjects/proxies in each group (observation vs video phase) who prefer comfort oriented care and who die in accordance with their stated preferences. | Measured on average within 48 hours of the palliative care service's referral of the subject to the research team, as well as 7-14 days, 2-3 months and 5-6 months post-discharge.

SECONDARY OUTCOMES:
The level of uncertainty regarding treatment preferences. | Measured on average within 48 hours of the palliative care service's referral of the subject to the research team.
Satisfaction with pain control and symptom management. | Measured on average within 48 hours of the palliative care service's referral of the subject to the research team, as well as 7-14 days, 2-3 months and 5-6 months post-discharge.
Healthcare proxy satisfaction with end-of-life care following subjects' death. | Measured at 7-14 days, 2-3 months or 5-6 months post-discharge.
Concordance between patient subjects' and staffs' ranking of symptoms. | Measured on average within 48 hours of the palliative care service's referral of the subject to the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paasche-Orlow, MD MA MPH, Principal Investigator — Boston University; Angelo Volandes, MD MPH, Principal Investigator — Massachusetts General Hospital; Nicole LaRue, MD, Study Director — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gillick MR. A broader role for advance medical planning. Ann Intern Med. 1995 Oct 15;123(8):621-4. doi: 10.7326/0003-4819-123-8-199510150-00009. PMID 7677304
- [Background] Emanuel LL, Barry MJ, Stoeckle JD, Ettelson LM, Emanuel EJ. Advance directives for medical care--a case for greater use. N Engl J Med. 1991 Mar 28;324(13):889-95. doi: 10.1056/NEJM199103283241305. PMID 2000111
- [Background] A controlled trial to improve care for seriously ill hospitalized patients. The study to understand prognoses and preferences for outcomes and risks of treatments (SUPPORT). The SUPPORT Principal Investigators. JAMA. 1995 Nov 22-29;274(20):1591-8. PMID 7474243
- [Background] Hofmann JC, Wenger NS, Davis RB, Teno J, Connors AF Jr, Desbiens N, Lynn J, Phillips RS. Patient preferences for communication with physicians about end-of-life decisions. SUPPORT Investigators. Study to Understand Prognoses and Preference for Outcomes and Risks of Treatment. Ann Intern Med. 1997 Jul 1;127(1):1-12. doi: 10.7326/0003-4819-127-1-199707010-00001. PMID 9214246
- [Background] Covinsky KE, Fuller JD, Yaffe K, Johnston CB, Hamel MB, Lynn J, Teno JM, Phillips RS. Communication and decision-making in seriously ill patients: findings of the SUPPORT project. The Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments. J Am Geriatr Soc. 2000 May;48(S1):S187-93. doi: 10.1111/j.1532-5415.2000.tb03131.x. PMID 10809474
- [Background] Garrett JM, Harris RP, Norburn JK, Patrick DL, Danis M. Life-sustaining treatments during terminal illness: who wants what? J Gen Intern Med. 1993 Jul;8(7):361-8. doi: 10.1007/BF02600073. PMID 8410396
- [Background] Forrow L. The green eggs and ham phenomena. Hastings Cent Rep. 1994 Nov-Dec;24(6):S29-32. No abstract available. PMID 7860277
- [Background] Tulsky JA, Fischer GS, Rose MR, Arnold RM. Opening the black box: how do physicians communicate about advance directives? Ann Intern Med. 1998 Sep 15;129(6):441-9. doi: 10.7326/0003-4819-129-6-199809150-00003. PMID 9735081
- [Background] Volandes AE, Paasche-Orlow MK, Barry MJ, Gillick MR, Minaker KL, Chang Y, Cook EF, Abbo ED, El-Jawahri A, Mitchell SL. Video decision support tool for advance care planning in dementia: randomised controlled trial. BMJ. 2009 May 28;338:b2159. doi: 10.1136/bmj.b2159. PMID 19477893
- [Background] Volandes AE, Barry MJ, Chang Y, Paasche-Orlow MK. Improving decision making at the end of life with video images. Med Decis Making. 2010 Jan-Feb;30(1):29-34. doi: 10.1177/0272989X09341587. Epub 2009 Aug 12. PMID 19675323
- [Background] El-Jawahri A, Podgurski LM, Eichler AF, Plotkin SR, Temel JS, Mitchell SL, Chang Y, Barry MJ, Volandes AE. Use of video to facilitate end-of-life discussions with patients with cancer: a randomized controlled trial. J Clin Oncol. 2010 Jan 10;28(2):305-10. doi: 10.1200/JCO.2009.24.7502. Epub 2009 Nov 30. PMID 19949010